CLINICAL TRIAL: NCT04914975
Title: The Effect of Neuromuscular Electrical Stimulation on Bowel Management in People with Chronic Spinal Cord Injury - a Pilot Study
Brief Title: The Effect of NMES on Bowel Management in People with Chronic SCI
Acronym: FES_Bowel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-27; 2021-00880 (Other: EKNZ)
Record Dates: First submitted 2021-05-31; First posted 2021-06-07 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Electric Stimulation Therapy; Bowel Dysfunction; Spinal Cord Injuries; Defecation Disorder
Keywords: Spinal Cord Injuries; Electrical Stimulation; Bowel Management; Transit Time; Incontinence; Quality of Life
MeSH Terms: conditions — Intestinal Diseases; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: repeated measures interventional single subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NMES Group (Experimental): Participants will receive neuromuscular electrical stimulation of the abdominal wall before defaecation for 30 minutes over the course of 16 weeks.
  Interventions: Other: Neuromuscular electrical stimulation

INTERVENTIONS:
Other: Neuromuscular electrical stimulation — The stimulation will be conducted at home or at the SPC for half an hour about 30 minutes before the usual bowel emptying time. Four adhesive electrodes are attached to the abdominal wall for the neuromuscular electrical stimulation. The abdominal muscles are stimulated in such a way that activation occurs, i.e. the muscle alternately contracts and relaxes again. The stimulation sessions will be documented with a defined protocol. In addition, the stool consistency is rated according to the Bristol Stool Form Scale.

SUMMARY:
It has been reported that 62% of all people with Spinal Cord Injury (SCI) have experienced faecal incontinence and that neurogenic bowel dysfunction (NBD) is a major sequela. As an alternative to abdominal massage or the use of suppositories, the electrical stimulation (ES) of the abdominal wall has been shown to be effective in decreasing the bowel transit time as well as decreasing constipation in children with slow-transit constipation. Due to the intrinsic nature of the guts' innervation, we expect to reproduce these positive effects in people with SCI through administration of neuromuscular electrical stimulation (NMES).

DETAILED DESCRIPTION:
A SCI entails devastating changes to a person's life. The extent of these changes depends on the level and degree of the lesion. NBD is one of the most important sequelae occurring in the majority of people with a SCI. It has been reported that 62% of people with SCI had experienced faecal incontinence . In fact, NBD is caused by a disruption of the autonomic nervous system leading to a disturbed colonic peristalsis. The enteric nervous system of the intestines is an intrinsic system that can function independently, but it is widely influenced by the autonomic nervous system. As such, its regulation is perturbed because the parasympathetic and the sympathetic nervous systems do modulate it but do not directly control the smooth muscle cells of the bowel . Depending on the level of the lesion, the bowel function can be affected in various ways ranging from constipation to overflow incontinence.

Hence, NBD has a major impact on the quality of life of paraplegics and tetraplegics. Not only is there a physical component to it consisting of constipation, haemorrhoids or abdominal distension but these gastrointestinal impairments also have a social aspect. People with SCI often end up avoiding social events and tend to isolate because of the fear of incontinence.

The immense expenditure of time for bowel evacuation is a consequence of the dyscoordination of faecal elimination. According to a survey study, 22% of all participants with SCI spend 31 to 60 minutes and 14% more than 60 minutes on bowel care per defecation. For example, people with an upper motor neuron lesion to their bowel are mainly confronted with faecal retention and constipation. Among the methods for bowel evacuation, the application of digital stimulation of the rectum and/or the insertion of a suppository are mostly used. Some people also use abdominal massage just before bowel evacuation . Only a few studies have investigated the effect of ES to the abdominal wall on the defaecation time in people with SCI and an upper motor neuron lesion but none investigated the defecation time in people with SCI with a lesion below the level of Th12. Nevertheless, the results of this therapeutic modality are very promising for different populations such as multiple sclerosis and children with slow-transit constipation by decreasing constipation and increasing transit times respectively.

By means of providing a more efficient and reliable method to support people with SCI in their bowel management strategy.A pilot study with a convenience sample of 20 out- and inpatients of the Swiss Paraplegic Centre will be conducted. Patients who have found a good bowel management method for themselves but claim to invest too much time in this routine are eligible for the study. During their participation, they should follow their usual routine after applying ES for 30 minutes before defaecation.

Based on the recent findings and clinical experience, it is hypothesized that NMES has the potential to reduce defaecation times as well as the bowel transit time in people with SCI experiencing NBD.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic and non-traumatic SCI; > 1 year
* Level of lesion: C2 - L5
* AIS score A/B/C/D
* Age: ≥ 18 years
* Urge to reduce defaecation time

Exclusion Criteria:

* Patients during primary rehabilitation
* Bladder stimulator
* Autonomic dysreflexia by application of ES of the abdominal wall
* Pregnancy: test in women of childbearing age (15 - 49 years)
* Opioid use
* Inflammatory bowel disease
* Cancerous tissue in abdominal region
* Patients' inability to follow the study, e.g. mental-health problems, language problems, dementia etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-04 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Neurogenic Bowel Dysfunction Score (NBDS) and the defaecation time from the stimulation protocol | 24 weeks
  Investigation of the effect of NMES on the change in defaecation time (minutes) and its relation to the change in NBDS between the follow-up visits and baseline

SECONDARY OUTCOMES:
Corn Test | 24 weeks; 5 time points
  "Corn Test" assessing bowel transit time
Bristol Stool Form Scale (BSFS) | 24 weeks; at each defaecation
  BSFS for stool consistency

OTHER OUTCOMES:
Qualiveen Short Form (SF) | 24 weeks; 5 times
  Qualiveen SF to assess bladder function
International Standards to document remaining Autonomic Function after Spinal Cord Injury (ISAFSCI) | 24 weeks; 5 times
  International Standards to document remaining Autonomic Function after Spinal Cord Injury (ISAFSCI)
Questionnaire of treatment effectiveness | 24 weeks; 2 times
  Questionnaire of treatment effectiveness containing 3 questions about the application of the stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Ines Bersch, PhD, Principal Investigator — International FES Centre - Swiss Paraplegic Centre Nottwil
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korsten MA, Fajardo NR, Rosman AS, Creasey GH, Spungen AM, Bauman WA. Difficulty with evacuation after spinal cord injury: colonic motility during sleep and effects of abdominal wall stimulation. J Rehabil Res Dev. 2004 Jan-Feb;41(1):95-100. doi: 10.1682/jrrd.2004.01.0095. PMID 15273902
- [Background] Krassioukov A, Eng JJ, Claxton G, Sakakibara BM, Shum S. Neurogenic bowel management after spinal cord injury: a systematic review of the evidence. Spinal Cord. 2010 Oct;48(10):718-33. doi: 10.1038/sc.2010.14. Epub 2010 Mar 9. PMID 20212501
- [Background] Clarke MC, Catto-Smith AG, King SK, Dinning PG, Cook IJ, Chase JW, Gibb SM, Robertson VJ, Di Simpson, Hutson JM, Southwell BR. Transabdominal electrical stimulation increases colonic propagating pressure waves in paediatric slow transit constipation. J Pediatr Surg. 2012 Dec;47(12):2279-84. doi: 10.1016/j.jpedsurg.2012.09.021. PMID 23217889
- [Background] Benevento BT, Sipski ML. Neurogenic bladder, neurogenic bowel, and sexual dysfunction in people with spinal cord injury. Phys Ther. 2002 Jun;82(6):601-12. PMID 12036401
- [Derived] Bersch I, Schafer K, Limacher A, Sonntag U, Baumberger M, Alberty M. The effect of neuromuscular electrical stimulation on bowel management in people with chronic spinal cord injury-An IDEAL 2a pilot study. Colorectal Dis. 2025 Nov;27(11):e70276. doi: 10.1111/codi.70276. PMID 41146588